CLINICAL TRIAL: NCT03455166
Title: Identification of New Prognostic Markers in Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BIO-ARP
Record Dates: First submitted 2017-12-05; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Psoriasis; Psoriatic Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psoriasis (Other)
  Interventions: Diagnostic Test: Serum Markers
- Psoriatic arthropathy (Other)
  Interventions: Diagnostic Test: Serum Markers

INTERVENTIONS:
Diagnostic Test: Serum Markers — Serum Markers

SUMMARY:
Identification of possible markers associated with the onset and / or progression of psoriatic arthritis through comparison in patients with psoriasis alone (Ps) and patients with psoriasis with joint involvement (PsA), plasma levels of a panel of cytokines referable to the Th17 pathway , together with serum levels of MMPs, TIMPs and markers of bone remodeling.

The primary objective of this study is to verify whether the arthropathy component has an effect on the metabolic activity of osteoblasts. This will be determined through the study of the differences in serum concentrations, between Ps and PsA subjects, of "CTx", the parameter best characterized in terms of analytical variability and intra- and inter-individual variability, in the field of bone metabolism.

The secondary objective is the verification of the differences in serum concentrations of the series of parameters specified above, in order to define a complete pattern of variations that can identify the molecular pathways involved in the definition of psoriatic arthropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* For Ps group:

plaque psoriasis no previous treatment with biological drugs

- For PsA group: plaque psoriasis with arthropathy no previous treatment with biological drugs but in treatment as per clinical practice or, alternatively, last treatment with drug suspended by a number of days double compared to the half-life of the drug

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Neoplasia in progress or previous (<5 years)
* Other acute or chronic inflammatory diseases
* Other rheumatological diseases
* Metabolic diseases of the primitive bone
* Recent bone fractures (<6 months)
* Anxiety, psychosis, depressive disorders
* Inability to understand the information provided by the recruiter doctor
* For Ps group:

treatment with biological drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Different markers concentration | 1 year
  Measurement in serum of: MMP-1, MMP-2, MMP-3, MMP-7, MMP-8, MMP-9, MMP-10, MMP-12, MMP-13, TIMP-1, TIMP-2, TIMP-3, TIMP-4, OPG, RANKL, PINP, CTx-I, DKK1, SOST,IL-1beta, IL-4, IL-6, IL-10, IL-17A, IL-17F, IL-21, IL-22, IL-23, IL-25, IL-31, IL-33, INFg, sCD40L, TNFalfa. Correlation with Ps or PsA, and with the severity of the disease

IPD SHARING:
Plan to Share IPD: No